CLINICAL TRIAL: NCT03157388
Title: The Effect of Gut Sterilisation on Macrophage Activation in Patients With Alcoholic Hepatitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1-10-72-1-15
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2018-12

CONDITIONS: Alcoholic Hepatitis
Keywords: inflammation; Macrophages; CD163
MeSH Terms: conditions — Hepatitis, Alcoholic; Inflammation | interventions — Gentamicins; Meropenem

STUDY DESIGN:
Intervention Model Description: 15 patients with alcoholic hepatitis will be consecutively included and compared to a historical cohort of AH patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Combined Vancomycin and Gentamycin and Meropenem
  Interventions: Drug: Combined Vancomycin and Gentamycin and Meropenem

INTERVENTIONS:
Drug: Combined Vancomycin and Gentamycin and Meropenem — The following combined antibiotic regime will be administered for eradication of gut bacteria.
  7 days combined antibiotic treatment, per oral route, once daily: vancomycin 500 mg (Vancomycin "Hospira"), powder for concentrate and gentamycin 40 mg ("Hexamycin®"), solution and meropenem 500 mg (Meropenem "Hospira"), powder for concentrate; The three drugs are dissolved and combined in approximately 100 ml of apple juice.

SUMMARY:
Alcoholic hepatitis (AH) is a severe alcohol induced hepatic inflammation that leads to jaundice and liver failure. Gut derived bacterial translocation to the liver is currently thought to be one of the main inflammatory drivers of the disease.

This project investigates the effects of gut sterilisation with broad spectrum antibiotics in patients with AH

DETAILED DESCRIPTION:
Alcoholic hepatitis (AH) is a severe alcohol induced hepatic inflammation that leads to jaundice and liver failure. The incidence of AH is increasing and the disease is associated with a high mortality. In spite of numerous clinical trials both treatment and prognosis have remained essentially unchanged for decades, emphasizing the need to improve our understanding of the disease mechanisms behind AH.

The current perception of the pathogenesis of alcohol-induced liver injury mainly derives from animal models, and the resident hepatic macrophages, the Kupffer cells, seem to play an important role. Activation of these cells may give rise to most of the hallmark clinical findings of AH: The cytokines released initiate hepatic inflammation and an acute phase response, recruit neutrophils, and activate stellate cells, contributing to the acute portal hypertension. Jaundice is due to intrahepatic cholestasis caused by down regulation of the bilirubin transporters on the basolateral hepatocyte membrane. Hepatic macrophages are thought to be activated by the bacterial derived endotoxins/lipopolysaccharides (LPS) present in the portal blood because of an alcohol-induced increase in gut-blood permeability with translocation of bacteria, as found in patients with alcoholic liver injury. LPS is recognized by the hepatic macrophages via a membrane complex including the pathogen recognition receptor molecule Toll-like receptor 4 (TLR-4). LPS Binding Proteins (LBP) produced by hepatocytes then bind and present LPS to the membrane glycoprotein CD14 that in turn activates TLR-4. In support of these mechanisms, alcohol-induced liver injury is reduced in knockout mice missing LBP, CD14, and TLR-4. Likewise, chemical destruction of hepatic macrophages in rats prevents alcohol-induced liver injury, as does cleansing the gut flora with antibiotics.

Human hepatic macrophages when activated, express their surface receptor CD163. We and others have previously shown that sCD163 is released from the liver in alcoholic liver disease, that its plasma concentration predicts mortality in patients with acute liver failure and is as a marker of portal hypertension and a predictor of clinical decompensation in patients with liver cirrhosis. Very recently we have directly demonstrated hepatic macrophage activation in human AH paralleling the disease severity, and to suggest this to be elicited by LPS.

The line of evidence presented above provides rationale for testing whether intervention toward bacterial translocation may result in a diminished immune response in human AH. Consequently, in this study the investigators seek to perform total gut microbiota eradication by combining 3 different orally administered antibiotics. The investigators have chosen antibiotics that are not absorbed into the systemic circulation, because the investigators want to limit the effects to the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

A first time diagnose of AH by a combination of physical and laboratory criteria:

1. A history of excessive alcohol ingestion (10 units or more per day) until at least three weeks before admission
2. Acute jaundice (developed over at most 2 weeks, serum bilirubin > 80 μmol/l).
3. liverbiopsy will be performed in case of doubt regarding the diagnosis.

Exclusion Criteria:

1. Non-native speaking Danish
2. Viral hepatitis,
3. Autoimmune liver disease,
4. Bile duct obstruction,
5. Liver tumours or any other cancer,
6. Presence of an infectious focus (either clinically assessed or based on chest x-ray, urine samples or ascites puncture),
7. On-going gastrointestinal bleeding or bleeding within the previous three months
8. Any prior immune-modulating therapy.
9. Any known gastrointestinal disease
10. Contraindications against/allergy towards the used antibiotics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Macrophage activation cd163 | 1 year
  Difference in serum levels of macrophage activation markers sCD163

SECONDARY OUTCOMES:
LBP | 1 year
  serum levels of Lipopolysaccaride binding protein
TNF alfa | 1 year
  serum levels of, Tumor Necrosis Factor-alfa
Interleukin-1b | 1 year
  serum levels of, Interleukin-1b

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik D Vilstrup, Professor, Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No